CLINICAL TRIAL: NCT04922671
Title: Towards Development of an Individualised Screening Tool By Utilising Cervical Length Measurement In Relation To Body Mass Index (BMI) For Early Identification And Intervention Of Preterm Birth
Brief Title: Development of a Screening Tool By Utilising Cervical Length Measurement In Relation To Body Mass Index (BMI) For Early Identification And Intervention Of Preterm Birth
Status: Completed | Type: Observational
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Nurul Iftida Binti Basri, Principal Investigator (Dr), Universiti Putra Malaysia
Other Study IDs: GM-IPM/2021/9695300
Record Dates: First submitted 2021-06-08; First posted 2021-06-10 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Cervical Length; Preterm Birth
Keywords: body mass index; preterm labour; preterm birth; cervical length
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective study where pregnant women between 16-24 weeks gestation attending the Antenatal Clinic, Fetomaternal clinic or Obstetrics & Gynaecology Admission Centre (OGAC) at Hospital Serdang or Hospital Pengajar UPM will be recruited. BMI will be taken both during booking of pregnancy and at recruitment. Cervical length will be measured via transvaginal scan at recruitment time. We aim to assess the association between body mass index, cervical length and risk of preterm birth.

DETAILED DESCRIPTION:
General Objective To assess the association between body mass index, cervical length and risk of preterm birth.

Specific Objectives

1. To examine the relationship between body mass index and cervical length
2. To identify cut-off value of cervical length leading to high risk of spontaneous preterm birth among Malaysian women
3. To assess the association between different cervical length and preterm birth
4. To examine the association between body mass index and preterm birth
5. To develop an individualised screening tool for assessing risk of preterm birth

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy between 16-24 weeks gestation
2. No history of previous spontaneous preterm birth (gestation between 24-36+6 weeks)
3. Agreement to follow up and consented for the study

Exclusion Criteria:

1. Major fetal anomaly
2. Multiple pregnancy
3. Uterine anatomic malformation
4. Those require iatrogenic preterm delivery due to various condition

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Antenatal women between 16-24 weeks gestation attending the Antenatal Clinic, Fetomaternal clinic or Obstetrics & Gynaecology Admission Centre (OGAC) at Hospital Serdang or Hospital Pengajar UPM
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
1. To examine the relationship between body mass index (BMI) and cervical length (CL) | till February 2023
  Association of BMI and CL
2. To identify cut-off value of cervical length | till February 2023
  Value leading to high risk of spontaneous preterm birth among Malaysian women
3. To assess the association between different cervical length and preterm birth | till February 2023
  Association of CL and PTB
4. To examine the association between body mass index and preterm birth | till February 2023
  Association of BMI and PTB
5. To develop an individualised screening tool for assessing risk of preterm birth | Till May 2023
  Attributable risk of preterm birth with relation to BMI and CL

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Hospital Pengajar UPM, Serdang, Selangor
  - Hospital Serdang, Serdang, Selangor

IPD SHARING:
Plan to Share IPD: No